CLINICAL TRIAL: NCT02079129
Title: A Novel Imaging Approach to Assess Paravalvular Leak for Transcatheter Valve Replacement
Brief Title: Paravalvular Leak for Transcatheter Valve Replacement
Acronym: PVL-TAVR
Status: Completed | Type: Observational
Sponsor: Baylor Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 013-185; PVL-TAVR (Other: Study Title)
Record Dates: First submitted 2014-03-03; First posted 2014-03-05 (Estimated); Last update posted 2020-01-22 (Actual); Status verified 2020-01

CONDITIONS: Paravalvular Leak; Transcatheter Valve Replacement
Keywords: agreement between cMRI PVL grading and TTE PVL grading; Edwards Sapien TAVR

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The study objective is to assess the agreement between cMRI PVL grading (based on regurgitant fraction) and TTE PVL grading (based on pressure half-time and the ratio of the jet arc to the circumference of the annulus).

DETAILED DESCRIPTION:
Background/Rationale

There are currently no objective, validated measures of paravalvular leak (PVL) by echocardiogram (Lerakis et al). The PARTNER 2 year outcomes demonstrated that even mild PVL is associated with poor prognosis (Kodali et al) and decreased survival after transaortic valve replacement (TAVR). It has been proposed that the severity of PVL could be measured based on a comparison of jet arc length and pressure half-time on color Doppler transthoracic echocardiogram (TTE) to the circumference of the valve annulus in the parasternal short-axis view. Accordingly, a jet arc corresponding to <10% of the annulus circumference indicates mild PVL, 10-20% moderate PVL, and >20% severe PVL. However, this grading method still needs to be validated against an independent reference standard such as Cardiac MRI (cMRI).

Cardiac MRI (cMRI) is a reliable way to measure PVL post-TAVR. It enables measurement of both regurgitant volume and regurgitant fraction using gradient echo-based phase-contrast sequence velocity flow mapping, accurately measuring forward stroke volume and backward regurgitant flow across the valve. Being independent of jet morphology, cMRI may be a superior way to follow patients post-TAVR. cMRI provides a quantitative assessment of the regurgitant fraction and can therefore serve as the reference standard for validation of TTE-based grading schemes.

Study Procedures

Patients seen at The Heart Hospital Baylor Plano (THHBP) will be enrolled into the study if they are eligible and provide written consent. Upon enrollment, demographic and clinical risk factors data will be collected for each patient. All patients will receive TTE and cMRI, within 1 week of each other, at their 30 days ± 14 days, 6 months ± 30 days, or 1 year ± 60 days follow up visit post-TAVR. TTE is usually performed at these follow-up visits as part of the routine clinical work up. All females of childbearing age will have a urine pregnancy test prior to cMRI. Patients will be assigned PVL severity grades according to the two diagnostic methods by Dr. Grayburn (TTEs), and Dr. Gopal (cMRIs). Both investigators will be blinded to each other grading results.

Risk/Benefit

MRI does not use ionizing radiation (high-energy radiation that can potentially cause damage to DNA, like the x-rays used CT scans).

There are no known harmful side-effects associated with temporary exposure to the strong magnetic field used by MRI scanners. However, there are important safety concerns to consider before performing or undergoing an MRI scan (U.S. Food and Drug Administration):

* The magnet may cause pacemakers, artificial limbs, and other implanted medical devices that contain metal to malfunction or heat up during the exam.
* Any loose metal object may cause damage or injury if it gets pulled toward the magnet.
* If a contrast agent is used, there is a slight risk of an allergic reaction. MRI contrast agents can cause problems in patients with significant kidney disease.
* Dyes from tattoos or tattooed eyeliner can cause skin or eye irritation.
* Medication patches can cause a skin burn.
* The wire leads used to monitor an electrocardiogram (ECG) trace or respiration during a scan must be placed carefully to avoid causing a skin burn.
* Prolonged exposure to radio waves during the scan could lead to slight warming of the body.

There are no known risks from a TTE. During this procedure, a technician obtains views of the heart by moving a transducer to different locations on the chest or abdominal wall. The transducer sends sound waves into the chest and picks up echoes that reflect off different parts of the heart (Cleveland Clinic).

Minimization of Risk

Patient safety during this study will be the highest priority. All diagnostic tests/treatments provided are commonly accepted and FDA approved. These test/treatments would be provided as part of the patients' post-operative follow up and the patients will not incur any additional health risks as subjects in this study. The patients will not incur any psychological, social, legal or economic risks by participating in this study.

Benefits

Subjects will not directly benefit from this research. The results of this study may provide important information for the medical imaging options for future valve replacement patients.

Adverse Events

Adverse Events (AEs) for purposes of this trial will include AEs related to TTE or MRI.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥18 years
* Patients eligible for implantation of Edwards Sapien aortic valve.

Exclusion Criteria:

* Pregnancy-Women of childbearing potential should have negative urine pregnancy test prior to enrollment
* Patients with implanted pacemaker
* Patients with implantable cardiac defibrillator
* Patients with contraindication to MRI
* Medically unable to provide consent
* Any surgical prosthesis
* Moderate or severe mitral regurgitation
* Central aortic valve leak

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study cohort will consist of 50 patients who have undergone Edwards Sapien TAVR who meet the following eligibility criteria and have provided written informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2014-01; Primary Completion 2018-07 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Assess the agreement between cMRI PVL grading (based on regurgitant fraction) and TTE PVL grading (based on pressure half-time and the ratio of the jet arc to the circumference of the annulus). | Up to 1 year +/- 60 days post TAVR.

CONTACTS AND LOCATIONS:
Overall Officials: Deepika Gopal, MD, Principal Investigator — Baylor Research Institute
Locations (1):
- The Heart Hospital Baylor, Plano, Texas, United States